CLINICAL TRIAL: NCT04437576
Title: Pregnancy and Latent Labor Biomarkers and Symptoms to Predict Cervical Dilation at Hospital Admission.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Bloomlife Technologies (Unknown); Medical Research Foundation, Oregon (Other); OHSU School of Nursing (Unknown)
Responsible Party: Principal Investigator, Ellen Tilden, Assistant Professor, Oregon Health and Science University
Other Study IDs: STUDY00020328
Record Dates: First submitted 2020-06-02; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Labor Onset Biomarkers; Labor Onset; Cervical Dilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed pilot investigation is a prospective, observational study of 300 healthy nulliparous women with spontaneous term labor onset. The specific aims of this study are to:

Aim #1: Characterize IL-8 (pro-inflammatory biomarker), basal body temperature, maternal heart rate, and electrical activity of the uterus prior to spontaneous onset of labor through the onset of active labor among nulliparous women. IL-8 will be quantified weekly, daily basal body temperature, as well as continuous maternal heart rate and electrical activity of the uterus throughout the transition from late pregnancy into active labor.

Aim #2: Characterize latent labor symptoms among nulliparous women in spontaneous labor. Using Likert scale, childbirth-specific, symptom-specific PROMIS measures,45 and open-ended questions will be quantified and characterize latent labor symptoms (e.g., intensity, frequency) and identify relevant themes.

Aim #3: Characterize trajectories of labor biomarkers and latent labor symptoms across latent labor duration. A modified growth mixture modeling approach to quantify subgroup phenotypes among nulliparous women in spontaneous latent labor will be employed.

Hypothesis 3.1. There will be significant congruence between higher biomarkers (e.g., higher IL-8, more uterine electrical activity) and symptoms that are more intense and frequent.

Hypothesis 3.2. At least two classes of laboring women with distinct trajectories of change in biomarkers and symptoms can be identified and will be associated with cervical dilation at hospital admission.

Exploratory Aim: Characterize biomarkers among nulliparous women with spontaneous labor onset vs. nulliparous women requiring labor induction for post-term gestation. Weekly IL-8, daily basal body temperature, as well as continuous maternal heart rate and electrical activity of the uterus throughout the transition from late pregnancy into active labor between those whose labor begins spontaneously and those whose labors are induced for post-term gestation will be quantified.

Exploratory Hypothesis. There will be different biomarker patterns between women with spontaneous labor onset vs. those without.

The Standard descriptive and inferential statistics as well as growth mixture modeling for quantitative aims will be used. The investigators will use thematic development for qualitative aims.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous
2. Maternal age of at least 20 years of age.
3. Maternal age of no greater than 39 years of age.
4. Viable, term pregnancy: ≥ 37 weeks gestation at time of signing study consent.
5. Able to understand and provide an informed consent.
6. Able to understand English.

Exclusion Criteria:

1. Multiple gestation (i.e., carrying >1 fetus)
2. Managing complex comorbidities (e.g., preeclampsia)
3. Documented fetal congenital anomalies
4. Preterm labor and birth
5. Persistent breech fetal position at term
6. Fetal death prior to the onset of labor
7. Any indication for planned cesarean birth (e.g., placenta previa)
8. Induction of labor for medical indication (e.g., oligohydramnios)

Ages: 20 Years to 39 Years | Sex: Female
Age Groups: Adult
Study Population: This is a study of reproductive age women 20-39 years of age being performed at Oregon Health & Science University (OHSU) in Portland, OR. It will include subjects who present for prenatal care in our outpatient Center for Women's Health Clinics and OHSU Labor and Delivery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Interleukin-8 (IL-8) expression during latent phase of labor to delivery | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Measure of IL-8 in serum
Changes in Basal body temperature during latent phase of labor to delivery | Daily from 37 weeks gestation until admission to hospital for labor
  Measure body temperature first thing every morning until admission to hospital for birth.
Change in Maternal heart rate during latent phase of labor to delivery | Continuously from 37 weeks gestation until admission to hospital for labor
  Wearable sensor worn to record heart rate continually.
Change in electrical activity of the uterus during latent phase of labor to delivery | Continuously from 37 weeks gestation until admission to hospital for labor
  Wearable sensor that records signals detected on the surface of the abdomen (e.g. signals generated by the uterus) and movements.

SECONDARY OUTCOMES:
Characterize latent labor symptoms among nulliparous women in spontaneous labor | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Quantify and characterize latent labor symptoms and identify relevant themes
Characterize trajectories of latent labor biomarkers across latent labor duration | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Quantify subgroup phenotypes among nulliparous women in spontaneous latent labor
Characterize trajectories of latent labor symptoms across latent labor duration | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Quantify subgroup phenotypes among nulliparous women in spontaneous latent labor using growth mixture modeling viewing longitudinal change.

OTHER OUTCOMES:
Change in Basal body temperature comparison in spontaneous labor vs induction | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Quantified weekly basal body temperature comparison throughout the transition from late pregnancy into active labor between those whose labor begins spontaneously and those whose labors are induced for post-term gestation.
Changes in continuous maternal heart rate comparison in spontaneous labor vs induction | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Quantified maternal heart rate comparison throughout the transition from late pregnancy into active labor between those whose labor begins spontaneously and those whose labors are induced for post-term gestation.
Changes in IL-8 comparison in spontaneous labor vs induction | week 37, week 38, week 39, week 40, week 41, week 42, upon admission for labor to OHSU
  Quantified weekly IL-8 comparison throughout the transition from late pregnancy into active labor between those whose labor begins spontaneously and those whose labors are induced for post-term gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Tilden, PhD, CNM, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No